CLINICAL TRIAL: NCT04586127
Title: Improving Care Coordination for Adolescents and Young Adults With Cancer: Implementing a Bridge Between Needs and Services
Brief Title: Improving Care Coordination for Adolescents and Young Adults With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00068240; P50CA244693 (NIH); P30CA012197 (NIH); 2T32CA122061 (NIH)
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Results first posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2022-07

CONDITIONS: Cancer
Keywords: adolescents; care coordination; cancer care needs
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescents and Young Adults Needs Assessment & Service Bridge (AYA NA-SB) (Experimental): Subjects will complete 2 online surveys over the course of 1 month; each should take about 15 minutes to complete.
  Interventions: Other: AYA NA-SB Questionnaire

INTERVENTIONS:
Other: AYA NA-SB Questionnaire — Questionnaire identifying cancer needs so that providers can connect subjects with services that might address them.

SUMMARY:
The purpose of this research is to test an intervention designed to identify cancer needs and connect patients with services that address those needs. Participation in this research will involve completing 2 online surveys over the course of 1 month; each should take about 15 minutes to complete.

DETAILED DESCRIPTION:
Adolescents and young Adults (AYA) Needs Assessment & Service Bridge (AYA NA-SB) includes a holistic Patient Reported Outcome Measures (PROM) assessing AYAs' physical, psychosocial and practical needs and a collection of referral pathways for connecting AYAs to services and resources based on the needs they report.

To assess the implementation of AYA NA-SB, the study team will pilot AYA NA-SB in the North Carolina Cancer Hospital (NCCH)/ UNC Children's Hospital, with a primary focus on implementation outcomes (i.e., feasibility, acceptability, appropriateness, fidelity). To establish proof-of-concept for AYA NA-SB, the study team will use pilot data to generate preliminary evidence on the extent to which AYA NA-SB addresses AYAs' reported needs.

ELIGIBILITY:
Inclusion Criteria:

* AYAs with cancer ages 18 through 39 currently undergoing cancer treatment at the North Carolina Cancer Hospital/ UNC Children's Hospital

Exclusion Criteria:

* Patients who decline to participate in the study

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Haines, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- North Carolina Cancer Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: In this single-arm feasibility pilot, the treatment arm completed the NA-SB Needs Assessment at baseline through a secure online survey platform, REDCap. The 57 items assessing AYAs' physical, psychosocial, practical need were preceded by items collecting demographic and clinical information from respondents. AYAs received a $15 incentive for completing the needs assessment. An AYA social worker or AYA nurse practitioner then reviewed their NA-SB Needs Assessment with them, addressed any needs that fell within their purview, and initiated referral pathways for any remaining needs. One month following completion of the NA-SB needs assessment, we engaged AYA pilot participants in an electronic postintervention survey assessing their perceptions of NA-SB and whether their needs were met. The postintervention survey was administered through REDCap and AYAs received a second $15 incentive for completing it.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 26
Completed | 21
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: young adults with cancer
Arm/Group | Treatment Arm
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 12
  Non-Hispanic Black | 9
  Hispanic (all races) | 1
  Non-Hispanic American Indian/Alaska Native | 1
  OTHER | 3
Cancer diagnosis [Count of Participants; unit: Participants]
  Leukemia | 9
  Breast | 3
  Cervical | 3
  Sarcoma | 3
  Male Reproductive | 2
  Non-Hodgkin Lymphoma | 1
  Hodgkin Lymphoma | 1
  Other female reproductive | 1
  Other | 3
Time since diagnosis [Count of Participants; unit: Participants]
  <3 months | 15
  3-6 months | 3
  7-12 months | 2
  >12 months | 6
Stage at diagnosis [Count of Participants; unit: Participants] — Participants self-reported cancer stage at diagnosis based on the information provided to them by their oncology care team. The "unknown/unstaged" option is for those who did not receive or remember receiving this information. Participants' respective physicians may have defined stages differently. In general, stage 0 is considered earliest/least advanced stage of cancer while stage IV describes most advanced cancer/ metastatic cancer. A higher stage represents more advanced cancer.
  Participants
    0 | 1
    I/II | 5
    III/IV | 5
    Unknown/ unstaged | 15
Insurance source [Count of Participants; unit: Participants]
  Employer/school | 10
  Spouse's employer/school | 1
  Parent | 2
  Medicaid | 6
  Medicare | 1
  Military/TRICARE | 1
  No insurance | 3
  Self-pay | 1
  Other | 1
Cohabitants [Count of Participants; unit: Participants]
  Lives alone | 2
  Parent(s) | 9
  Sibling(s) | 1
  Spouse/partner | 9
  Roommate(s) | 4
  Other | 1
School status [Count of Participants; unit: Participants]
  In school | 7
  Not in school | 19
Working status [Count of Participants; unit: Participants]
  Working | 13
  Not working | 13

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Intervention Measure (FIM) AYA
Description: Questionnaire measuring the extent to which AYA NA-SB can be successfully used in cancer programs. Score ranges from 1 to 5 with higher score denoting higher feasibility.
Time Frame: Week 5
Population: young adults with cancer
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 21
units on a scale | 4.52 (0.50)

2. Primary Outcome: Acceptability of Intervention Measure (AIM) AYA
Description: Questionnaire measuring perception of whether AYA-NA-SB is agreeable, palatable, or satisfactory to users. Score ranges from 1 to 5 with a higher score denoting higher acceptability.
Time Frame: Week 12
Population: young adults with cancer
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 21
units on a scale | 4.5 (0.5)

3. Primary Outcome: Intervention Appropriateness Measure (IAM) AYA
Description: Questionnaire measuring perception of AYA-NA-SB's fit, relevance, or compatibility with the context in which it will be used. Score ranges from 1 to 5 with a higher score denoting higher appropriateness
Time Frame: Week 5
Population: young adults with cancer
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 21
units on a scale | 4.4 (0.489)

4. Primary Outcome: Number of Participants Who Received Services
Description: Care coordination will be assessed by the proportion of Adolescents and Young Adults (AYAs) who reported needs who received services from across disciplines to address reported needs within one month of needs assessment completion.
Time Frame: Week 12
Population: young adults with cancer who reported needs
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 16
Participants | 13

5. Primary Outcome: Needs Met Questionnaire
Description: Questionnaire assessing, among AYAs who reported needs and reported receiving follow-up care, AYAs' perception of the degree to which their needs were adequately addressed during the study period. Scores range from 1 to 5 where higher scores denote that needs were met.
Time Frame: Week 12
Population: young adults with cancer who reported needs and reported receiving follow-up care
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 13
units on a scale | 3.7 (1.6)

6. Secondary Outcome: Number of AYA Needs
Description: Average number of needs reported by AYAs.
Time Frame: Week 12
Population: young adults with cancer
Measure: Mean (Inter-Quartile Range); unit: needs reported
Arm/Group | Treatment Arm
Number analyzed (Participants) | 26
needs reported | 13 [2 to 21]

ADVERSE EVENTS:
Time Frame: from baseline up through 14 months
Description: clinicaltrials.gov definition
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 1/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT04586127/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT04586127/ICF_000.pdf